CLINICAL TRIAL: NCT02276586
Title: Prospective Clinical Evaluation of Periodontal Response to Different Prosthetic Margin Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova, School of Dental Medicine (Other)
Responsible Party: Principal Investigator, Eriberto Bressan, Chairman, Department of Periodontology, University of Padova, School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2737P
Record Dates: First submitted 2014-10-09; First posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Gingival Recession; Gingival Disease; Gingival Bleeding
MeSH Terms: conditions — Gingival Recession; Gingival Diseases; Gingival Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Horizontal Tooth preparation
  Interventions: Procedure: Horizontal Tooth preparation
- Group 2 (Experimental): Vertical tooth preparation
  Interventions: Procedure: Vertical Tooth preparation

INTERVENTIONS:
Procedure: Horizontal Tooth preparation — Round parallel chamfer diamond burs were used for teeth preparation; coarse first (151 micron) and extra-fine after (25 micron)
  Arms: Group 1
Procedure: Vertical Tooth preparation — Long flame diamond burs were used for teeth preparation; coarse first (151 micron) and extra-fine after (25 micron)
  Arms: Group 2

SUMMARY:
Background: The actual literature is consistent in considering potential negative effects of sub-gingival prosthetic margins on the periodontal health, but no research has focused the attention on the type of prosthetic margin designs. Hence, the aim of the present study is to evaluate if a horizontal finishing line (deep chamfer preparation) may have a different influence on periodontal soft tissue in comparison with a vertical finishing line (feather edge preparation).

Methods: A prospective randomized controlled double blind clinical trial with one single operator and three experienced examiners was performed. One hundred and six crowns were prepared with horizontal tooth preparation while ninety-four with vertical tooth preparation. All the margins were positioned within the periodontal sulcus, at 0.5mm sub-gingivally and all the all-ceramic restorations were cemented with resin cement. Periodontal Probing Depth (PPD), Plaque Index (PI), Gingival Index (GI) and Gingival Bleeding on Probing (BOP) were recorded prior to tooth preparation and twelve month after crown cementation. Also, at 12 months follow-up, the gingival margin position was related to the crown margin position.

ELIGIBILITY:
Inclusion Criteria:

The patient inclusion criteria were as follows:

1. dentate patients treatment planned for single unit restorations in the esthetic zone (from 1st premolar forward)
2. periodontal probing depth prior to tooth preparation ≤4mm, with no bleeding on probing and no plaque
3. >30 years of age
4. full mouth plaque score (FMPS) and full mouth bleeding scores (FMBS) <20% at study baseline
5. eventual loss of attachment limited only to areas different from the sites included in the study.

The patient exclusion criteria were as follows:

1. patient with medical history in which any dental intervention would be contraindicated
2. any local or systemic disease, condition or medication that might compromise healing and affect the periodontium
3. dental caries or periodontal disease in the remaining teeth
4. inability or unwillingness to return for follow-up visit.

Exlusion Criteria:

1. patients with systemic diseases (such as heart, coagulation, and leukocyte diseases or metabolic disorders)
2. history of radiation therapy in the head and neck region within 12 months prior to surgical phase
3. current treatment with steroids
4. neurological or psychiatric condition that could interfere with good oral hygiene
5. immunocompromised status, including infection with human immunodeficiency virus
6. smoking habit (more than 10 cigarettes/day)
7. drug or alcohol abuse
8. inadequate compliance
9. patients who received bone regeneration procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Plaque Index (PI) | Change from Baseline Plaque Index at 12 months post intervention
  Plaque Index (PI), according to Silness & Loe
Periodontal Probing Depth (PPD) | Change from Baseline Periodontal Probing Depth (PPD) at 12 months post intervention
  Periodontal Probing Depth (PPD) measured at three different facial sites (mesial, facial, distal), with the utilization of a periodontal probe (UNC periodontal probe, Hu-Friedy, Chicago, IL) recording the measurements to the nearest millimeter.
Gingival Index (GI) | Change from Baseline Gingival Index (GI) at 12 months post intervention
  Gingival Index (GI), according to Silness & Loe
Bleeding on Probing (BOP) | Change from Baseline Bleeding on Probing (BOP) at 12 months post intervention
  Bleeding on Probing (BOP), according to Ainamo & Bay (presence or absence)
Gingival recession (GR) | Change from Baseline Gingival recession (GR) at 12 months post intervention
  Gingival margin position related to the crown margin

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Padua, PD, Italy